CLINICAL TRIAL: NCT00477594
Title: An Open-Label Extension Study to Assess the Long-term Safety and Efficacy of Mipomersen in Subjects With Familial Hypercholesterolemia
Brief Title: Open Label Extension of ISIS 301012 (Mipomersen) to Treat Familial Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 301012-CS17; 2007-001024-12 (EudraCT Number)
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Results first posted 2013-04-05 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Lipid Metabolism, Inborn Errors; Hypercholesterolemia, Autosomal Dominant; Hyperlipidemias; Metabolic Diseases; Hyperlipoproteinemia Type II; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Metabolic Disorder; Congenital Abnormalities; Hypercholesterolemia; Hyperlipoproteinemias; Dyslipidemias; Lipid Metabolism Disorders
Keywords: Familial Hypercholesterolemia; Heterozygous Familial Hypercholesterolemia; Homozygous Familial Hypercholesterolemia; ISIS 301012; mipomersen; Open Label Extension
MeSH Terms: conditions — Lipid Metabolism, Inborn Errors; Hyperlipoproteinemia Type II; Hyperlipidemias; Metabolic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Congenital Abnormalities; Hypercholesterolemia; Hyperlipoproteinemias; Dyslipidemias; Lipid Metabolism Disorders; Homozygous Familial Hypercholesterolemia | interventions — mipomersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mipomersen 200 mg per week (Experimental): Participants received 200 mg mipomersen once a week by subcutaneous injection, for up to 3 years.
  Interventions: Drug: mipomersen sodium
- Mipomersen 200 mg every other week (Experimental): Participants received 200 mg mipomersen every other week by subcutaneous injection, for up to 3 years. Participants could receive mipomersen 200 mg once a week at the Investigator's discretion after the first 52 weeks of the treatment period.
  Interventions: Drug: mipomersen sodium

INTERVENTIONS:
Drug: mipomersen sodium — 200 mg/ml, in 1 ml solution for subcutaneous injection.
  Other Names: ISIS 301012; Kynamro™

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of extended dosing of mipomersen in patients with familial hypercholesterolemia on lipid-lowering therapy who have completed either the 301012-CS8 (NCT00280995) or 301012-CS9 (NCT00281008) clinical drug trials.

DETAILED DESCRIPTION:
Familial Hypercholesterolemia (FH) is an autosomal dominant metabolic disorder characterized by markedly elevated low density lipoprotein (LDL), premature onset of atherosclerosis, and development of xanthomata. There are two distinct subpopulations that have a high unmet medical need due to the lack of alternative therapy: homozygotes, who have two defective LDL receptor (LDL-R) genes, and heterozygotes with a history of cardiovascular disease (CVD) on maximally tolerated therapy. Treatment for FH is directed at lowering plasma levels of LDL-C.

Mipomersen is an antisense drug targeted to human apolipoprotein B (apoB), the principal apolipoprotein of atherogenic LDL-C and its metabolic precursor, very low density lipoprotein (VLDL). Mipomersen is complimentary to the coding region of the messenger ribonucleic acid (mRNA) for apo-B. Inhibition of apo-B would be expected to impair VLDL synthesis and result in lowered levels of LDL-C.

In early clinical trials, mipomersen has been shown to reduce levels of LDL-C to recommended target levels in some participants.

This was an open-label extension study, which consisted of a ≤2-week screening period, up to 3 years of treatment with mipomersen, and a 24-week post-treatment follow-up period. Patients who participated in Cohorts A, B, or C in study 301012-CS9 were randomized in a 1:1 ratio to mipomersen 200 mg once a week (QW) or 200 mg mipomersen every other week (QOW) for up to 3 years. Patients randomized to mipomersen 200 mg QOW were allowed to receive mipomersen 200 mg QW at the Investigator's discretion after the first 52 weeks of the treatment period. Patients who participated in study 301012-CS8 or Cohort D of study 301012-CS9 received 200 mg mipomersen QW for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

- Satisfactory completion of dosing and Week 7 or Week 15 assessments (depending on the treatment and dose received) in their initial study (Protocol 301012-CS8 (NCT00280995) or 301012-CS9 (NCT00281008)).

Exclusion Criteria:

- Have a new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with patient's participation in or completion of the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-05; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (5):
- United States (5):
  - Chicago, Illinois
  - Auburn, Maine
  - Biddeford, Maine
  - Scarborough, Maine
  - Cincinnati, Ohio

REFERENCES:
- [Derived] Patel N, Hegele RA. Mipomersen as a potential adjunctive therapy for hypercholesterolemia. Expert Opin Pharmacother. 2010 Oct;11(15):2569-72. doi: 10.1517/14656566.2010.512006. PMID 20707601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who completed dosing in study 301012-CS8 (NCT00280995) or 301012-CS9 (NCT00281008) at a site in the U.S. with an acceptable safety profile, per Investigator judgment, were eligible to enroll in this study.
Pre-assignment Details: Patients who participated in Cohorts A, B, or C in study 301012-CS9 were randomized in a 1:1 ratio to mipomersen 200 mg once a week (QW) or 200 mg mipomersen every other week (QOW). Patients who participated in study 301012-CS8 or Cohort D of study 301012-CS9 received 200 mg mipomersen QW.
Period: Year 1 and Year 2
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Started | 16 | 5
Completed | 7 | 1
Not Completed | 9 | 4
Not completed — Adverse Event | 4 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 1 | 0
Period: Year 3
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Started | 4 | 0
Completed | 2 | 0
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Follow-up Period
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Started | 16 | 5
Completed | 13 | 4
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week | Total
Number analyzed (Participants) | 16 | 5 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (11.6) | 54.6 (15.7) | 48.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 12 | 3 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 5 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  White | 14 | 5 | 19
  Other race | 1 | 0 | 1
  Multiple | 1 | 0 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (5.60) | 27.4 (4.81) | 28.6 (5.34)
Metabolic syndrome [Number; unit: participants] — A patient was classified as having metabolic syndrome if any 3 of the following risk factors existed: 1) Waist circumference ≥102 cm (men) or ≥88 cm (women); 2) Triglycerides ≥150 mg/dL*; 3) High density lipoprotein cholesterol <40 mg/dL (men) or <50 mg/dL (women)*; 4) Systolic blood pressure ≥130 or diastolic ≥85 mmHg*; 5) Fasting glucose ≥100 mg/dL*.
  * = or on medication for the specified risk factor.
  participants
    No | 8 | 3 | 11
    Yes | 8 | 2 | 10
Tobacco Use [Number; unit: participants]
  Current | 1 | 0 | 1
  Non-current | 5 | 2 | 7
  Never | 10 | 3 | 13
Alcohol use [Number; unit: participants]
  Current | 13 | 3 | 16
  Non-current | 1 | 0 | 1
  Never | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: LDL cholesterol was measured in mg/dL. Samples were taken following an overnight fast. For patients with triglycerides <400 mg/dL, LDL-C was obtained using Friedewald's calculation; and for patients with triglycerides ≥400 mg/dL, LDL-C was directly measured by the central laboratory using ultracentrifugation. For patients who were on placebo in the index study or who took their last dose of mipomersen ≥6 months prior to first dose in this study, Baseline is defined as the last measurement prior to first dose in this study. For participants who took their last dose of mipomersen less than 6 months before starting this study, Baseline is defined as the last measurement taken prior to receiving a first dose in the index study.
Time Frame: Baseline and Weeks 52 and 104
Population: The Safety Set included all enrolled patients who received at least 1 injection of study drug. "N" indicates the number of participants with available data at the specified time point.
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Week 52 [N=13, 4] | -16.2 [-41.8 to -7.8] | -2.6 [-10.2 to 14.8]
  Week 104 [N=7, 1] | -32.4 [-38.8 to -16.6] | 30.6 [30.6 to 30.6]
  Week 104/Early Termination [N=16, 5] | -13.8 [-31.4 to -3.0] | 9.5 [3.4 to 11.5]

2. Primary Outcome: Low-density Lipoprotein Cholesterol (LDL-C) Over Time
Description: Samples were taken following an overnight fast. For patients with triglycerides <400 mg/dL, LDL-C was obtained using Friedewald's calculation; and for patients with triglycerides ≥400 mg/dL, LDL-C was directly measured by the central laboratory using ultracentrifugation. For patients who were on placebo in the index study or who took their last dose of mipomersen ≥6 months prior to first dose in this study, Baseline is defined as the last measurement prior to first dose in this study. For participants who took their last dose of mipomersen less than 6 months before starting this study, Baseline is defined as the last measurement taken prior to receiving a first dose in the index study.
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
mg/dL
  Baseline [N=16, 5] | 177 [134 to 205] | 131 [124 to 147]
  Week 52 [N=13, 4] | 145 [106 to 173] | 127 [124 to 139]
  Week 104 [N=7, 1] | 121 [82 to 156] | 162 [162 to 162]
  Week 104/Early Termination [N=16, 5} | 144 [116 to 213] | 161 [146 to 162]

3. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B
Description: Apolipoprotein B was measured in mg/dL. Samples were taken following an overnight fast. For patients who were on placebo in the index study or who took their last dose of mipomersen ≥6 months prior to first dose in this study, Baseline is defined as the last measurement prior to first dose in this study. For participants who took their last dose of mipomersen less than 6 months before starting this study, Baseline is defined as the last measurement taken prior to receiving a first dose in the index study.
Time Frame: Baseline and Weeks 52 and 104
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Week 52 [N=13, 4] | -25.9 [-39.1 to -11.0] | -7.3 [-19.7 to 7.7]
  Week 104 [N=7, 1] | -27.2 [-39.7 to -22.4] | 20.8 [20.8 to 20.8]
  Week 104/Early Termination [N=16, 5] | -15.8 [-26.2 to -3.5] | -3.7 [-14.9 to -1.6]

4. Secondary Outcome: Apolipoprotein B Over Time
Description: For patients who were on placebo in the index study or who took their last dose of mipomersen ≥6 months prior to first dose in this study, Baseline is defined as the last measurement prior to first dose in this study. For participants who took their last dose of mipomersen less than 6 months before starting this study, Baseline is defined as the last measurement taken prior to receiving a first dose in the index study.
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
mg/dL
  Baseline [N=16, 5] | 148 [127 to 181] | 124 [109 to 154]
  Week 52 [N=13, 4] | 136 [102 to 146] | 110 [104 to 123]
  Week 104 [N=7, 1] | 110 [73 to 146] | 128 [128 to 128]
  Week 104/Early Termination [N=16, 5] | 132 [104 to 175] | 128 [122 to 131]

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol
Description: Total cholesterol was measured in mg/dL. Samples were taken following an overnight fast.
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Week 52 [N=13, 4] | -10.5 [-26.8 to -6.4] | -6.5 [-13.4 to 8.6]
  Week 104 [N=7, 1] | -25.3 [-29.2 to -18.0] | -1.5 [-1.5 to -1.5]
  Week 104/Early Termination [N=16, 5] | -11.2 [-24.2 to -2.4] | -1.5 [-1.7 to 2.6]

6. Secondary Outcome: Total Cholesterol Over Time
Description: as for outcome 4
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
mg/dL
  Baseline [N=16, 5] | 251 [206 to 293] | 233 [199 to 235]
  Week 52 [N=13, 4] | 216 [173 to 245] | 203 [192 to 220]
  Week 104 [N=7, 1] | 209 [143 to 209] | 196 [196 to 196]
  Week 104/Early Termination [N=16, 5] | 209 [193 to 297] | 231 [199 to 239]

7. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol
Description: Non-high-density lipoprotein cholesterol was measured in mg/dL. Samples were taken following an overnight fast.
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Week 52 [N=13, 4] | -24.7 [-40.5 to -12.6] | -6.7 [-15.0 to 9.5]
  Week 104 [N=7, 1] | -34.3 [-37.9 to -21.6] | 17.2 [17.2 to 17.2]
  Week 104/Early Termination [N=16, 5] | -16.5 [-31.2 to -6.6] | 3.7 [-3.0 to 14.1]

8. Secondary Outcome: Non-High-Density Lipoprotein Cholesterol Over Time
Description: as for outcome 4
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
mg/dL
  Baseline [N=16, 5] | 206 [167 to 253] | 151 [149 to 203]
  Week 52 [N=13, 4] | 167 [134 to 208] | 150 [140 to 164]
  Week 104 [N=7, 1] | 161 [95 to 174] | 177 [177 to 177]
  Week 104/Early Termination [N=16, 5] | 164 [151 to 255] | 177 [170 to 197]

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: AEs were considered as related if assessed by the Investigator as possibly, probably or definitely related to study drug. The severity of each event was assessed using the following categories: Mild (symptom(s) barely noticeable to the patient or do not make the patient uncomfortable); Moderate (symptom(s) of a sufficient severity to make the patient uncomfortable, performance of daily activities is influenced) or Severe (symptom(s) of a sufficient severity to cause the patient severe discomfort, may cause cessation of treatment with the study drug). Serious AEs (SAEs) are those that resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in an important medical event that may have jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: 2 years
Population: Safety set
Measure: Number; unit: participants
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
participants
  Any adverse event | 16 | 5
  Treatment-related adverse event | 16 | 5
  Mild adverse event | 5 | 2
  Moderate adverse event | 8 | 3
  Severe adverse event | 3 | 0
  Serious adverse event | 4 | 2
  Adverse event leading to treatment discontinuation | 4 | 2

10. Secondary Outcome: Percent Change From Baseline in Clinical Chemistry Parameters
Time Frame: Baseline and Week 104 or the Early Termination visit for participants who did not complete 2 years of treatment.
Population: Safety set.
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Alanine aminotransferase (ALT) | 63.73 (112.98) | 29.96 (80.01)
  Aspartate aminotransferase (AST) | 48.73 (86.00) | 3.53 (39.14)
  Bilirubin, Indirect | 13.81 (20.56) | 12.50 (29.86)
  Bilirubin, Total | 34.79 (57.97) | 0.48 (10.96)
  Blood Urea Nitrogen (BUN) | 6.08 (22.90) | -11.06 (16.56)
  Creatine Kinase | -17.24 (36.85) | 40.95 (149.95)
  Creatinine | -9.94 (12.54) | -9.84 (14.05)
  Glomerular Filtration Rate (GFR) | 16.20 (24.56) | 15.49 (21.58)

11. Secondary Outcome: Percent Change From Baseline in Hematology Parameters
Time Frame: Baseline and Week 104 or the Early Termination visit for participants who did not complete 2 years of treatment
Population: Safety set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Hematocrit | -0.04 (8.69) | -5.24 (3.69)
  Hemoglobin | 0.90 (7.61) | -4.24 (4.44)
  Leukocytes | -0.80 (31.95) | -5.99 (43.17)
  Platelets | -8.55 (11.88) | -1.36 (12.31)

12. Secondary Outcome: Percent Change From Baseline in Blood Pressure
Time Frame: Baseline and Week 104 or the Early Termination visit for participants who did not complete 2 years of treatment.
Population: Safety set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Systolic Blood Pressure | 6.99 (12.33) | 2.35 (12.54)
  Diastolic Blood Pressure | -0.88 (11.31) | 10.67 (15.35)

13. Secondary Outcome: Percent Change From Baseline in Pulse Rate
Time Frame: Baseline and Week 104 or the Early Termination visit for participants who did not complete 2 years of treatment.
Population: Safety set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline | 4.89 (14.41) | 6.28 (17.45)

14. Secondary Outcome: Percent Change From Baseline in Respiratory Rate
Time Frame: Baseline and Week 104 or the Early Termination visit for participants who did not complete 2 years of treatment.
Population: Safety set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline | 0.87 (10.57) | -4.44 (13.30)

15. Other Pre Specified Outcome: Percent Change From Baseline in Triglycerides
Description: Triglycerides were measured in mg/dL. Samples were taken following an overnight fast.
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Week 52 [N=13, 4] | -30.2 [-36.3 to -26.7] | -27.0 [-43.0 to -3.1]
  Week 104 [N=7, 1] | -46.8 [-58.2 to -30.2] | -44.8 [-44.8 to -44.8]
  Week 104/Early Termination [N=16, 5] | -34.3 [-42.9 to 2.2] | -34.7 [-36.1 to 9.0]

16. Other Pre Specified Outcome: Triglycerides Over Time
Description: as for outcome 4
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
mg/dL
  Baseline [N=16, 5] | 167 [96 to 254] | 134 [92 to 199]
  Week 52 [N=13, 4] | 102 [67 to 150] | 90 [80 to 123]
  Week 104 [N=7, 1] | 77 [67 to 113] | 74 [74 to 74]
  Week 104/Early Termination [N=16, 5] | 98 [76 to 180] | 122 [97 to 130]

17. Other Pre Specified Outcome: Percent Change From Baseline in Lipoprotein(a)
Description: Lipoprotein(a) was measured in mg/dL. Samples were taken following an overnight fast.
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Week 52 [N=13, 4] | -20.2 [-34.3 to -4.7] | 0.0 [-27.3 to 0.0]
  Week 104 [N=7, 1] | -30.7 [-32.7 to -24.1] | 0.0 [0.0 to 0.0]
  Week 104/Early Termination [N=16, 5] | -18.2 [-31.0 to 0.0] | -20.0 [-25.0 to 0.0]

18. Other Pre Specified Outcome: Lipoprotein(a) Over Time
Description: as for outcome 4
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
mg/dL
  Baseline [N=16, 5] | 50 [15 to 98] | 5 [3 to 11]
  Week 52 [N=13, 4] | 54 [23 to 75] | 4 [3 to 5]
  Week 104 [N=7, 1] | 49 [33 to 79] | 3 [3 to 3]
  Week 104/Early Termination [N=16, 5] | 47 [24 to 71] | 4 [3 to 4]

19. Other Pre Specified Outcome: Percent Change From Baseline in Very-Low-Density Lipoprotein (VLDL) Cholesterol
Description: Very-Low-Density Lipoprotein (VLDL) Cholesterol was measured in mg/dL. Samples were taken following an overnight fast.
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Week 52 [N=13, 4] | -31.6 [-37.1 to -25.0] | -25.9 [-43.6 to -2.8]
  Week 104 [N=7, 1] | -48.6 [-58.3 to -31.6] | -44.4 [-44.4 to -44.4]
  Week 104/Early Termination [N=16, 5] | -34.0 [-44.0 to 2.8] | -35.0 [-35.7 to 5.6]

20. Other Pre Specified Outcome: Very-Low-Density Lipoprotein (VLDL) Cholesterol Over Time
Description: as for outcome 4
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
mg/dL
  Baseline [N=16, 5] | 34 [19 to 51] | 27 [18 to 40]
  Week 52 [N=13, 4] | 20 [13 to 30] | 18 [16 to 25]
  Week 104 [N=7, 1] | 15 [13 to 23] | 15 [15 to 15]
  Week 104/Early Termination [N=16, 5] | 20 [15 to 36] | 24 [19 to 26]

21. Other Pre Specified Outcome: Percent Change From Baseline in Ratio of Low-density Lipoprotein Cholesterol to High-density Lipoprotein Cholesterol
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Week 52 [N=13, 4] | -33.5 [-43.6 to -25.8] | 2.6 [-11.8 to 10.2]
  Week 104 [N=7, 1] | -41.2 [-57.8 to -34.6] | 230.1 [230.1 to 230.1]
  Week 104/Early Termination [N=16, 5] | -24.9 [-38.2 to -18.5] | 15.2 [3.1 to 35.7]

22. Other Pre Specified Outcome: Ratio of Low-density Lipoprotein Cholesterol to High-density Lipoprotein Cholesterol Over Time
Description: as for outcome 4
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
ratio
  Baseline [N=16, 5] | 4 [3 to 6] | 3 [2 to 4]
  Week 52 [N=13, 4] | 3 [2 to 4] | 3 [2 to 3]
  Week 104 [N=7, 1] | 3 [2 to 4] | 9 [9 to 9]
  Week 104/Early Termination [N=16, 5] | 3 [2 to 4] | 5 [2 to 5]

23. Other Pre Specified Outcome: Percent Change From Baseline in Apolipoprotein A1
Description: Apolipoprotein A1 was measured in mg/dL. Samples were taken following an overnight fast.
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Week 52 [N=13, 4] | 4.6 [-4.3 to 11.2] | 7.4 [-5.3 to 17.0]
  Week 104 [N=7, 1] | 5.9 [-2.7 to 7.6] | -55.1 [-55.1 to -55.1]
  Week 104/Early Termination [N=16, 5] | 6.3 [-0.7 to 9.5] | -7.9 [-11.8 to -3.4]

24. Other Pre Specified Outcome: Apolipoprotein A1 Over Time
Description: as for outcome 4
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
mg/dL
  Baseline [N=16, 5] | 132 [120 to 149] | 149 [147 to 178]
  Week 52 [N=13, 4] | 139 [123 to 160] | 159 [144 to 178]
  Week 104 [N=7, 1] | 142 [113 to 155] | 66 [66 to 66]
  Week 104/Early Termination [N=16, 5] | 141 [129 to 153] | 144 [126 to 164]

25. Other Pre Specified Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol
Description: High-Density Lipoprotein (HDL) Cholesterol was measured in mg/dL. Samples were taken following an overnight fast.
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
percentage of baseline
  Week 52 [N=13, 4] | 12.8 [6.4 to 32.4] | 6.8 [-4.9 to 12.0]
  Week 104 [N=7, 1] | 14.9 [6.1 to 43.8] | -60.4 [-60.4 to -60.4]
  Week 104/Early Termination [N=16, 5] | 15.3 [4.9 to 26.9] | -17.9 [-19.6 to 6.3]

26. Other Pre Specified Outcome: High-Density Lipoprotein Cholesterol Over Time
Description: as for outcome 4
Time Frame: Baseline and Weeks 52 and 104.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Number analyzed (Participants) | 16 | 5
mg/dL
  Baseline [N=16, 5] | 40 [33 to 46] | 52 [48 to 56]
  Week 52 [N=13, 4] | 46 [41 to 50] | 54 [43 to 66]
  Week 104 [N=7, 1] | 47 [35 to 48] | 19 [19 to 19]
  Week 104/Early Termination [N=16, 5] | 47 [40 to 50] | 45 [34 to 58]

ADVERSE EVENTS:
Time Frame: Up to 3 years.
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Mipomersen 200 mg Per Week | Mipomersen 200 mg Every Other Week
Serious Adverse Events (participants affected / at risk) | 4/16 | 3/5
Other Adverse Events (participants affected / at risk) | 16/16 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mipomersen 200 mg Per Week (N=16) | Mipomersen 200 mg Every Other Week (N=5)
Angina pectoris (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mipomersen 200 mg Per Week (N=16) | Mipomersen 200 mg Every Other Week (N=5)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 2
Cardiomegaly (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Thyroid cyst (Endocrine disorders) | 1 | 0
Arcus lipoides (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 2
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Adverse drug reaction (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Feeling jittery (General disorders) | 0 | 1
Influenza like illness (General disorders) | 2 | 3
Injection site anaesthesia (General disorders) | 1 | 0
Injection site coldness (General disorders) | 1 | 0
Injection site discolouration (General disorders) | 3 | 1
Injection site erythema (General disorders) | 10 | 2
Injection site haematoma (General disorders) | 1 | 3
Injection site haemorrhage (General disorders) | 2 | 0
Injection site hypertrophy (General disorders) | 2 | 0
Injection site pain (General disorders) | 3 | 2
Injection site pruritus (General disorders) | 2 | 2
Injection site rash (General disorders) | 1 | 0
Injection site reaction (General disorders) | 7 | 1
Injection site swelling (General disorders) | 1 | 2
Injection site urticaria (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Acarodermatitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0
Splinter (Injury, poisoning and procedural complications) | 0 | 1
Wrong technique in drug usage process (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 5 | 0
Platelet count decreased (Investigations) | 1 | 0
Protein urine present (Investigations) | 2 | 0
Urine analysis abnormal (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Grief reaction (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 12 months after completion of the study the PI may publish the results of his/her data from the study. The PI shall provide the sponsor with an advance copy at least 60 days prior to planned submission and the Sponsor shall have 60 days to review (contracts have variable timeframes; maximum times are stated here). The sponsor may request the deletion of any confidential information, or a delay in submission for an additional period not to exceed 90 days.